CLINICAL TRIAL: NCT01968655
Title: Expanded Access to B-Domain Deleted Recombinant Porcine Factor VIII (OBI-1) in the Treatment of Acquired Hemophilia A Due to Factor VIII Inhibitory Auto-antibodies
Status: No longer available | Type: Expanded Access
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: OBI-1-301a
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Acquired Hemophilia A
Keywords: Factor VIII Inhibitory Auto-antibodies
MeSH Terms: conditions — Factor 8 deficiency, acquired

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: OBI-1 — OBI-1 is a B domain deleted recombinant porcine factor VIII
  Other Names: B-Domain Deleted Recombinant Porcine Factor VIII

SUMMARY:
To provide emergency access to OBI-1 for patients with Acquired Hemophilia and a serious bleeding episode who do not have access to an active clinical study site associated with the OBI-1-301 study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from participant or their legal representative.
* Participants with acquired hemophilia with autoimmune inhibitors to human factor VIII.
* Has a serious bleeding episode, as documented by the investigator.
* Be willing and able to follow all instructions and attend all study visits.
* Participants taking anti-thrombotics may be included depending on the time elapsed since taking such medications.
* Life expectancy of at least 90 days prior to the onset of the bleeding episode.

Exclusion Criteria:

* Hemodynamically unstable after blood transfusion, fluid resuscitation and pharmacologic or volume replacement pressor therapy.
* Has an established reason for bleeding that is not correctable.
* Bleeding episode assessed likely to resolve on its own if left untreated.
* Anti-OBI-1 inhibitor that exceeds 20 BU (prospectively or retrospectively).
* Subsequent bleeding episode at the site of the initial qualifying bleeding episode within 2 weeks following the final OBI-1 dose for the initial qualifying bleeding episode, or subsequent bleeding episode at a different site than the initial qualifying bleeding episode within 1 week following the final OBI-1 dose for the initial qualifying bleeding episode will not be considered "new" qualifying bleeding episodes.
* Prior history of bleeding disorder other than acquired hemophilia.
* Known major sensitivity (anaphylactoid reactions) to pig or hamster products.
* Use of hemophilia medication within 3 to 6 (depending on medication) hours prior to OBI-1 administration.
* Participation in any other clinical study within 30 days of the first OBI 1 treatment.
* Anticipated need for treatment or device during the study that may interfere with the evaluation.
* Abnormal baseline findings
* Inability or unwillingness to comply with the study design, protocol requirements, or the follow-up procedures.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (4):
  - National Institutes of Health Warren G. Magnuson Clinical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Penn State, Hershey, Pennsylvania
  - Vanderbilt Hemostasis/Hemophilia Clinic, Nashville, Tennessee